CLINICAL TRIAL: NCT01909271
Title: Tailored Approaches to Stroke Health Education
Acronym: TASHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Chief of Staff of Neurology Associate Professor of Clinical Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAK5853; 1U54NS081765-01 (NIH)
Record Dates: First submitted 2013-07-22; First posted 2013-07-26 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Community Health Education; Minority Health; healthcare disparities
MeSH Terms: conditions — Stroke; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive education through a novel program called Stroke Education Film Viewing.
  Interventions: Behavioral: Stroke Education Film Viewing
- Usual Care Group (Other): Participants will receive education through Stroke Education Pamphlet Exposure.
  Interventions: Other: Stroke Education Pamphlet Exposure

INTERVENTIONS:
Behavioral: Stroke Education Film Viewing — A novel, culturally tailored intervention using storytelling (narrative persuasion) in the form of two professionally produced 12-min films (in English and Spanish), in minority populations in New York City.
  Arms: Intervention Group
Other: Stroke Education Pamphlet Exposure — "Usual Care": Stroke Education pamphlet and brochure distribution.
  Arms: Usual Care Group

SUMMARY:
The overarching goal of the proposed intervention is to reduce stroke disparities by overcoming pre-hospital barriers related to emergency stroke treatment and facilitating the appropriate response to acute stroke using a novel culturally-tailored and sustainable approach developed by an experienced transdisciplinary team. Building on our previous work, in which the investigators have identified barriers to increasing stroke literacy and behavioral intent to call 911, the investigators will develop and evaluate the effectiveness of a novel, culturally tailored intervention using storytelling (narrative persuasion) in the form of two professionally produced 12-minute films (in English and Spanish), in minority populations in New York City (NYC). Behavioral intent to call 911 will be assessed immediately after viewing the film, 6 months later, and one year later.

DETAILED DESCRIPTION:
Stroke is the leading cause of adult disability and costs U.S. taxpayers >$60 billion annually. Interventions designed to educate patients to seek treatment sooner when a stroke occurs may increase low rates of treatment with thrombolysis (current rates 3% national average). Thrombolysis can increase the odds of minimal to zero disability from stroke if emergency medical system response times and in-hospital response times are optimized (maximum time from symptom onset to intravenous thrombolysis is 4.5 hours). Black and Hispanic Americans have higher stroke incidence compared to Whites and are less likely to receive thrombolysis for acute stroke. The latency to hospital arrival is largely dependent on patients' recognition of stroke symptoms, and immediate presentation to the emergency department. The investigators have found very low stroke literacy rates among Blacks and Hispanics compared to Whites, which may, in part, be responsible for disparities in acute stroke treatment.

ELIGIBILITY:
Inclusion Criteria:

1. No prior history of stroke;
2. High risk (defined as a history of one or more stroke risk factor (hypertension (HTN), diabetes, tobacco, abdominal obesity, heart disease, high cholesterol);
3. Over age 34 years at onset of intervention (we have selected this age cut off due to the large increase in stroke incidence among minority groups at age 34 );
4. Self-identified as Black or Hispanic; and
5. Member of a church congregation who lives in a household with a telephone.

Exclusion Criteria:

1. Participant is unable to give consent;
2. A modified Rankin score > 4 at baseline;
3. history of dementia; and
4. terminal illness, or other medical illness resulting in mortality < 1 year.

Min Age: 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Score on Stroke Action Test | Within one hour of stroke education intervention.
  The Stroke Action Test (STAT) contains 21 items that name or describe stroke symptoms from all 5 groups of warning signs and 7 items that are nonstroke symptoms. For each item, the respondent selects 1 of 4 options: call 911, call doctor, wait 1 hour, or wait 1 day. For scoring purposes, each correct response receives 1 point; incorrect responses receive 0 points. The total score is reported as percent of correct responses. Scores range from 0% to 100% with a higher score indicating a better outcome.

SECONDARY OUTCOMES:
Score on Stroke Action Test | Within six months of stroke education intervention.
  The Stroke Action Test (STAT) contains 21 items that name or describe stroke symptoms from all 5 groups of warning signs and 7 items that are nonstroke symptoms. For each item, the respondent selects 1 of 4 options: call 911, call doctor, wait 1 hour, or wait 1 day. For scoring purposes, each correct response receives 1 point; incorrect responses receive 0 points. The total score is reported as percent of correct responses. Scores range from 0% to 100% with a higher score indicating a better outcome.
Score on Stroke Action Test | Within one year of stroke education intervention.
  The Stroke Action Test (STAT) contains 21 items that name or describe stroke symptoms from all 5 groups of warning signs and 7 items that are nonstroke symptoms. For each item, the respondent selects 1 of 4 options: call 911, call doctor, wait 1 hour, or wait 1 day. For scoring purposes, each correct response receives 1 point; incorrect responses receive 0 points. The total score is reported as percent of correct responses. Scores range from 0% to 100% with a higher score indicating a better outcome.

OTHER OUTCOMES:
Time to emergency room after suffering a stroke | Up to 3.5 years post-intervention
  This measures the time in getting to the emergency room after having suffered a stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Olajide. A Williams, MD, MS, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, Neurological Institute, New York, New York
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams O, Teresi J, Eimicke JP, Abel-Bey A, Hassankhani M, Valdez L, Gomez Chan L, Kong J, Ramirez M, Ravenell J, Ogedegbe G, Noble JM. Effect of Stroke Education Pamphlets vs a 12-Minute Culturally Tailored Stroke Film on Stroke Preparedness Among Black and Hispanic Churchgoers: A Cluster Randomized Clinical Trial. JAMA Neurol. 2019 Oct 1;76(10):1211-1218. doi: 10.1001/jamaneurol.2019.1741. PMID 31260028
- [Derived] Ravenell J, Leighton-Herrmann E, Abel-Bey A, DeSorbo A, Teresi J, Valdez L, Gordillo M, Gerin W, Hecht M, Ramirez M, Noble J, Cohn E, Jean-Louis G, Spruill T, Waddy S, Ogedegbe G, Williams O. Tailored approaches to stroke health education (TASHE): study protocol for a randomized controlled trial. Trials. 2015 Apr 19;16:176. doi: 10.1186/s13063-015-0703-4. PMID 25927452